CLINICAL TRIAL: NCT00909051
Title: Diabetes Treatment by Glucobay® With a Special Therapeutic View to Chosen Patient Groups
Brief Title: GlucoVIP - Diabetes Treatment by Glucobay® With a Special Therapeutic View to Chosen Patient Groups
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14284; GB0701 (Other: Company internal)
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Acarbose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Acarbose (Glucobay, BAYG5421)

INTERVENTIONS:
Drug: Acarbose (Glucobay, BAYG5421) — Patients with diabetes type 2 newly treated with Glucobay

SUMMARY:
Evaluation of safety and effectiveness of Glucobay® under daily-life treatment conditions in a large sample of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with untreated or pretreated diabetes mellitus or patients for which acarbose is indicated and without acarbose treatment within the last three months before study inclusion. The decision for treatment type and duration is taken by the investigator and is made before inclusion into the study.

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with untreated or pretreated diabetes mellitus type 2
  * No Glucobay® intake within the last 3 months before documentation of initial visit
  * Exclusion Criteria: contraindication stated in the local Glucobay® product information; warnings and precautions must be considered.
Sampling Method: Non-Probability Sample
Enrollment: 15729 (Actual)
Dates: Start 2009-03-24 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2010-12-31 (Actual)

PRIMARY OUTCOMES:
Data collection on patients weight and waist circumference, fasting blood glucose, postprandial blood glucose (2h), HbA1C; exploratory analysis according to patient groups (concomitant cardiovascular disease groups, BMI) | During observation period of three months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (16):
- Multiple Locations, Algeria
- Multiple Locations, Bosnia and Herzegovina
- Multiple Locations, Cambodia
- Multiple Locations, China
- Multiple Locations, Hong Kong
- Multiple Locations, India
- Multiple Locations, Indonesia
- Multiple Locations, Malaysia
- Multiple Locations, Moldova
- Multiple Locations, Pakistan
- Multiple Locations, Philippines
- Multiple Locations, Russia
- Multiple Locations, Singapore
- Multiple Locations, South Korea
- Multiple Locations, Thailand
- Multiple Locations, Vietnam

REFERENCES:
- [Result] Zhang W, Kim D, Philip E, Miyan Z, Barykina I, Schmidt B, Stein H; Gluco VIP study. A multinational, observational study to investigate the efficacy, safety and tolerability of acarbose as add-on or monotherapy in a range of patients: the Gluco VIP study. Clin Drug Investig. 2013 Apr;33(4):263-74. doi: 10.1007/s40261-013-0063-3. PMID 23435929